CLINICAL TRIAL: NCT00140348
Title: A Phase I/II Dose Escalation and Efficacy Trial of GVAX® Prostate Cancer Vaccine in Patients With Metastatic Hormone-Refractory Prostate Cancer
Brief Title: Dose Escalation and Efficacy Trial of GVAX® Prostate Cancer Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-0010
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Advanced Prostate Cancer; Metastatic; Hormone-refractory; GVAX; Vaccine; Allogeneic cells
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Biological: Immunotherapy allogeneic GM-CSF secreting cellular vaccine

SUMMARY:
The purpose of this study is to evaluate clinical and laboratory safety in patients receiving 4 different doses of GVAX® Prostate Cancer Vaccine in order to determine a maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the prostate
* Metastatic prostate cancer deemed to be unresponsive or refractory to hormone therapy
* Detectable metastases
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Transitional cell, small cell, neuroendocrine, or squamous cell prostate cancer
* Significant cancer related pain
* Prior gene therapy, chemotherapy, or immunotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2001-12; Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - South Orange County Medical Research Center, Laguna Woods, California
  - UCSF, San Francisco, California
  - West Coast Clinical Research, Tarzana, California
  - South Florida Medical Research, Aventura, Florida
  - Emory University, Atlanta, Georgia
  - Carle Cancer Center, Urbana, Illinois
  - Northeast Indiana Research, Fort Wayne, Indiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Fox Chase cancer Center, Philadelphia, Pennsylvania
  - Urology San Antonio, San Antonio, Texas
  - Virginia Mason Med. Crt., Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington